CLINICAL TRIAL: NCT04612491
Title: Effect of Pre-operative Consultation on Patient Anxiety and Satisfaction Following First-time Mohs Micrographic Surgery
Brief Title: Pre-operative Consultation on Patient Anxiety and First-time Mohs Micrographic Surgery
Status: Terminated | Type: Observational
Why Stopped: Closure Requested by Cancer Center for Slow Accrual
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1094298
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-06

CONDITIONS: Anxiety; Surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-operative Consultation
  Interventions: Behavioral: Pre-operative Consultation
- No consultation

INTERVENTIONS:
Behavioral: Pre-operative Consultation — Pre-operative consultation will be given before Mohs surgery
  Groups: Pre-operative Consultation

SUMMARY:
To determine if in-office pre-operative consultation has a significant effect on the anxiety level and overall post-operative satisfaction of patients undergoing first time Mohs surgery

DETAILED DESCRIPTION:
This study is designed to determine if having a seperate in-office pre-operative consultation with the dermatologist before having a dermatologic procedure has any effect on patient anxiety levels and satisfaction following the procedure. The goal of the study is to help us understand if pre-operative consultation is beneficial to patients to reduce anxiety and increase satisfaction following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or older

  * Able to provide consent for participation
  * Fluency in English
  * Presenting for first-time Mohs surgery for treatment of a cutaneous malignancy

Exclusion Criteria:

* • Patients under 18 years old

  * Prisoners
  * Patients unable to provide consent
  * History of prior Mohs surgery
  * Patients requiring multi-disciplinary care (i.e. Involvement of other surgical specialties such as Plastic Surgery or Ophthalmology for reconstruction)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at r the UC Davis Dermatology Clinic who are scheduled for the Mohs procedure.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
The score on the PSQ-18 survey following the Mohs procedure | 2 years
  The PSQ-18 (aka patient satisfaction questionaire-18) is a validated assessment tool developed to measure holistic patient satisfaction with the aspects of clinical care (assessing six domains of patient satisfaction: technical quality, interpersonal manner, communication, financial aspects of care, accessibility of care and time spent with the physician), and by virtue of its brevity (18 questions taking an average of 3-4 minutes to complete) has great utility for measuring patient satisfaction in the clinical setting. Each question ranges from 1-5. Lower scores are better.
  The primary null hypothesis for this study is that mean PSQ-18 survey scores do not differ between patients receiving pre-operative consultation versus those not receiving this intervention.

SECONDARY OUTCOMES:
Patient anxiety as measured on the 10-point VAS scale for anxiety | 2 years
  The VAS is a horizontal line with a scale ranging from "no anxiety at all" to "extremely anxious." By measuring the position of the patient's response on the line, a score out of 10 will be generated. The VAS for anxiety will be administered to enrolled patients at three time points: randomization (consent visit), pre-operatively on day of Mohs surgery and post-operatively on the day of the Mohs surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No